CLINICAL TRIAL: NCT06348823
Title: Relationship Between Soft Tissue Volume and Gingival Phenotype: a Novel Classification System
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Collaborators: British University In Egypt (Other)
Responsible Party: Principal Investigator, ahmed hamdy mahmoud, assistant lecturer, British University In Egypt
Other Study IDs: BritishUE
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-04

CONDITIONS: Gingival Biotype; Soft Tissue
Keywords: soft tissue volume

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- thin biotype group: All subjects received oral hygiene instructions and, if needed, a dental cleaning of plaque and calculus. After calibration using digital photographs, intraoral scans, and CBCT, one dentist, who was not involved in the screening phase to avoid any bias, obtained all clinical parameters (gingival biotype, probing depth, gingival thickness, gingival width). Two test subjects were examined prior starting with enrollment and data collection.
  Interventions: Diagnostic Test: volume survey
- thick biotype group: All subjects received oral hygiene instructions and, if needed, a dental cleaning of plaque and calculus. After calibration using digital photographs, intraoral scans, and CBCT, one dentist, who was not involved in the screening phase to avoid any bias, obtained all clinical parameters (gingival biotype, probing depth, gingival thickness, gingival width). Two test subjects were examined prior starting with enrollment and data collection.
  Interventions: Diagnostic Test: volume survey

INTERVENTIONS:
Diagnostic Test: volume survey — All subjects received oral hygiene instructions and, if needed, a dental cleaning of plaque and calculus. After calibration using digital photographs, intraoral scans, and CBCT, one dentist, who was not involved in the screening phase to avoid any bias, obtained all clinical parameters (gingival biotype, probing depth, gingival thickness, gingival width). Two test subjects were examined prior starting with enrollment and data collection.

SUMMARY:
Different classifications to describe alveolar ridge defects have been published over the past years but no single classification has been developed concerning soft tissue volume around teeth or dental implants. Moreover, while several studies investigated the effect of various augmentation techniques and materials on soft tissue volume change and volume stability there is a real gap of knowledge regarding how to evaluate the available soft tissue volume and when to consider it sufficient or deficient which would definitely improve clinical decision making and treatment planing. Therefore, our primary aim was to assess the application of a novel classification system based on the correlation between buccal soft tissue volume and gingival biotypes and, also to assess the sensitivity of such novel method.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients in a healthy systemic condition who required comprehensive dental treatment.
2. Both genders with age group > 18 years old.
3. CBCT scans will be obtained as a part of the comprehensive dental treatment.
4. Patients should approve to deliver a signature to a written consent after study nature explanation.

Exclusion Criteria:

1. Patients with severe smoking habits >10 cig \ day.
2. Pregnant females, decisional impaired individuals, Prisoners and handicapped patients.
3. Patients having poor oral hygiene or not wanting to carry out oral hygiene measures.
4. Patients with fillings or crowns in the central incisors.
5. Patients on any medication affecting the soft tissue health (e.g., amlodipine, Cyclosporine A, hydantoin),

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cross sectional observational clinical study will include ---- patients that will be recruited from the outpatient clinic of the department of Oral Medicine, Periodontology, and Diagnosis, Faculty of Dentistry, The British University in Egypt.
  Demographic data of all patients will be collected. Patients will be clearly instructed about the purpose of this study and will give their consent by signing an informed consent.
  The study will be started after being accepted by the faculty of Dentistry, The British University in Egypt Research Ethics Committee. The study tracks the guideline of the research ethical committee in line with the Helsinki Declaration of 1975.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2024-02-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
soft tissue volume - biotype correlation | 3 months
  The association between gingival biotype and buccal soft tissue volume will be analyzed. Sensitivity and specificity of this novel method will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED HAMDY MAHMOUD MAHMOUD, Principal Investigator — British University In Egypt
Locations (1):
- Ahmed Hamdy, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided